CLINICAL TRIAL: NCT01010113
Title: Growth of Infants Consuming Starter Formula Containing Synbiotics
Brief Title: Effects of a Synbiotics-containing Starter Formula on Infant Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09.02 INF
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Infant Nutrition
Keywords: infants; prebiotics; probiotics; safety
MeSH Terms: interventions — Prebiotics; Infant Formula; Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test formula 1 (Placebo Comparator): Standard formula with prebiotics
  Interventions: Other: Standard infant formula with prebiotics
- test product (Experimental): Infant formula with synbiotics
  Interventions: Other: Infant formula with synbiotics

INTERVENTIONS:
Other: Standard infant formula with prebiotics — From 0-6 months of age. As per standard requirement
  Arms: Test formula 1
Other: Infant formula with synbiotics — From 0-6 months of age as per standard requirement
  Arms: test product

SUMMARY:
In this study the investigators want to evaluate the satiety of two infant formulas, one containing prebiotics and the other containing synbiotics. Rate of weight gain, a proxy measurement for the healthy development of an infant, will be assessed in both groups and compared to the growth observed in the WHO Child Growth Standards in order to demonstrate non inferiority.

DETAILED DESCRIPTION:
Growth studies continue to be a centrepiece of clinical evaluation of infant formulas. In order to standardize growth, the investigator proposes to calculate the weight-for-age Z-score related to the WHO Child Growth Standards. Z-scores express the difference between the measurement of an individual and the median value of the reference population as a proportion of the SD of the reference population taking into account age and gender.

The hypothesis to be tested is that infants fed with starter formula with prebiotics and probiotics blend and those fed only with probiotics will grow as much as infants in the reference growth of WHO.

Other parameters such as digestive tolerance, frequency of morbidity and microbiota pattern will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Age at point of enrolment ≤14 days
* Birthweight ≥2500g and ≤4500g
* Full term infant ≥37 weeks gestation and ≤42 weeks gestation
* Singleton births
* Having obtained his/her or his/her legal representative's informed consent

Exclusion Criteria:

* Congenital illness or malformation that may affect normal growth
* Significant pre-natal or post-natal disease
* Re-hospitalisation for more than 2 days during the first 14 days of life (Exceptionally, infants hospitalized because of jaundice may be enrolled in the study.)
* Receiving infant formula containing probiotics and/or prebiotics prior to enrollment and/or at the time of enrollment
* Patient who cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial prior to the beginning of this study

Ages: 11 Days to 17 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
mean weight gain | 6 months

SECONDARY OUTCOMES:
digestive tolerance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lee Le Ye, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Lee le Y, Bharani R, Biswas A, Lee J, Tran LA, Pecquet S, Steenhout P. Normal growth of infants receiving an infant formula containing Lactobacillus reuteri, galacto-oligosaccharides, and fructo-oligosaccharide: a randomized controlled trial. Matern Health Neonatol Perinatol. 2015 Apr 7;1:9. doi: 10.1186/s40748-015-0008-3. eCollection 2015. PMID 27057326